CLINICAL TRIAL: NCT05831566
Title: Expertise Asthma COPD Program with Digital Support
Acronym: EXACT@home
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Franciscus Gasthuis (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Hans in 't Veen, Principal investigator, Franciscus Gasthuis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL79996.100.22
Record Dates: First submitted 2022-12-20; First posted 2023-04-26 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Asthma
Keywords: severe asthma; ehealth; digital home monitoring; difficult to treat asthma; treatable traits; assessment; biologics
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Open-label, randomized controlled trial with a superiority design. Patients will be randomly assigned to one of two groups in parallel for the duration of the study. They will either recieve biologics directly or they will undergo an in-dept assessment to map the asthma diagnosis in more detail.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (EXACT@home) (Experimental): These patients will first undergo the systematic assessment (=EXACT@home) of +/- 6 weeks including a systematic anamnesis, questionnaires and home monitoring with multiple digital devices (digital inhaler, activity tracker, hand-held spirometer and FeNO measuring device) and a Personal Digital Health Environment (PDHE). Based on this evaluation and the degree of asthma control a treatment will be chosen: optimization of treatable traits if present and/or biologics.
  The personal digital healthcare environment and digital inhaler will be used for 12 months and the activity tracker, hand-held spirometer and FeNO measuring device will be used for 12 weeks.
  Interventions: Drug: Budesonide/Formoterol fumarate dihydrate
- Control arm (biologics) (Active Comparator): These patients will immediately receive a biologic after the indication is determined at the regional asthma Multi-Disciplinary Team Meeting (MDTM). These patients also have access to the Personal Digital Health Environment (PDHE) and they will also use the digital inhaler but without being able to see their own results or receiving feedback/reminders (silent).
  The personal digital healthcare environment and digital inhaler will be used for 12 months.
  Interventions: Drug: Budesonide/Formoterol fumarate dihydrate

INTERVENTIONS:
Drug: Budesonide/Formoterol fumarate dihydrate — The Digihaler will measure use of inhalation medication and inhaler technique and will give feedback and reminders. The aim is to improve adherence en inhaler technique. The device/medicinal product will be used for 12 months.
  It will be used in both groups, but patients in the intervention group are not able to see their own results and will not receive feedback/reminders.
  Other Names: Budesonide Formoterol (BF) Digihaler Digital System (DS)

SUMMARY:
The aim EXACT@Home is to create an evidence-based health program using e.g. questionnaires, a digital health platform and multiple digital devices to further improve the assessment of patients diagnosed with severe asthma. By better charting treatable traits (e.g. poor adherence, physical inactivity, dysfunctional breathing), we expect to improve the indication for the use of biologics. One the devices that will be used is also a medicinal product: a digital inhaler, which monitors adherence and inhaler technique through its connected application and aims to improve adherence and inhaler technique with reminders and notifications. Next to this an activity tracker, hand-held spirometer and FeNO measuring device will be used. The information of the devices will be collected in a Personal Digital Healthcare Environment (PDHE). Patients diagnosed with severe asthma according to the regional asthma Multi-Disciplinary Team Meeting (MDTM) eligible for a treatment with biologics will be included. Half of the patients will immediately receive a biologic. The other half will first undergo the systematic assessment including home monitoring (=EXACT@home) and afterwards a treatment will be chosen based on this evaluation: optimization of treatable traits when present and/or biologics. The chosen treatment of both, the intervention and control group, will be evaluated during 11-12 months.

DETAILED DESCRIPTION:
Rationale:

Asthma is a common multifactorial disease with chronic inflammation of the lower airways, which is in most cases adequately treated by inhalation medication. 17% of asthma patients have difficult-to-treat asthma, which is uncontrolled despite of an optimal treatment with medication due to the presence of 'treatable traits'. Examples of treatable traits are poor adherence to ICS/LABA therapy and inhaler technique, dysfunctional breathing, physical inactivity and behavior. Severe and refractory asthma is a subtype of difficult-to-treat asthma and only occurs if the asthma is uncontrolled despite optimized treatment with medication and addressing of treatable traits, which occurs in only 3.7% of all asthma patients. This group of patients is responsible for a high burden of overall disease, as well as large healthcare costs.Treatment options with biologics have fundamentally changed the care for patients with severe asthma by giving a relevant improvement in asthma control, the number of asthma exacerbations and quality of life. On the other hand, these drugs are also very expensive and must be given for the correct indication.

The Centre of Excellence for severe Asthma, Franciscus Gasthuis & Vlietland, Rotterdam organizes a weekly Multi-Disciplinary Team Meeting (MDTM) for hospitals in the South-West of the Netherlands to discuss their patients with problematic asthma and to start a treatment with biologics approved for severe asthma (in this document further called biologics). Despite maximal efforts of all stakeholders, the complete overview of a patient and the treatable traits is often hampered by the complexity and heterogeneity of severe asthma.

The aim of the EXACT@Home (Expertise Asthma COPD program with digital support) study is to further improve the assessment of treatable traits using ehealth before considering treatment with biologics.

Objectives:

Primary objective: To investigate if the EXACT@home program results in a reduced percentage of patients treated with biologics by means of systematically targeting treatable traits measured after 6 months of follow up.

Secondary objectives: To determine whether the use of EXACT@home results in a reduced percentage of patients treated with biologicals after 11-12 months. Next to this it will be investigated if EXACT@home has an influence on quality of life, asthma control, dyspnea perception, lung function, exacerbation frequency, prednisolone use, direct healthcare consumption, self-management skills, patient satisfaction, adherence to ICS/LABA therapy and inhaler technique, physical activity, sleep and vital parameters. Next to this, breath pattern analysis will be performed with the electronic nose (eNose). Moreover, the safety of the Digital inhaler (BF-Digihaler-DS from Teva) and eNose (Spironose from Breathomix) and the course of the treatment in each patient will also be investigated.

Study design:

Open-label, randomized controlled trial with a superiority design.

Study population:

Patients aged ≥ 18 years, in which the diagnosis severe and refractory asthma and eligibility for treatment with biologics was determined at the regional asthma MDTM will be asked to participate in this project.

Intervention (if applicable):

Patients will be randomized in 2 groups (intervention - and control group). The intervention group participates in a holistic assessment called EXACT@home consisting of a period of 6 weeks addressing diagnosis, asthma phenotype and treatable traits using e.g. questionnaires and digital devices measuring airway obstruction, eosinophilic airway inflammation, adherence to ICS/LABA therapy, inhalation technique, movement, vital parameters and sleep. The information of the devices and all other information concerning the patient will be stored in an 'Personal Digital Healthcare Environment (PDHE)'. Afterwards the collected data will be evaluated. Based on this evaluation and the degree of asthma control the type of treatment will be determined: optimization of 'treatable traits' or start of treatment with biologics. The control group will immediately start the treatment with biologics. The chosen treatment of both, the intervention and control group, will be evaluated during 11-12 months.

Main study parameters/endpoints:

Study parameter primary outcome:

Difference between the intervention and control group in the percentage of patients treated with biologicals after 6 months of follow up.

Study parameters secondary outcome:

The percentage of patients treated with biologicals after 11-12 months of follow up, quality of life, asthma control, dyspnea perception, lung function, exacerbation frequency, prednisolone use, direct healthcare consumption, self-management skills, patient satisfaction, adherence to ICS/LABA therapy, inhaler technique, physical activity, slap, vital parameters, breath pattern analysis with the eNose, safety of the digital inhaler and eNose and the course of the treatment in each patient.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The possible burden of the intervention group is temporarily postponing an effective treatment with biologics in favour of in depth extensive assessment in patients with a severe disease for a short period of at least 6 weeks. On the other hand, the patient could benefit from the EXACT@home assessment possibly leading to a personalized treatment, in which a treatment with biologics might not be necessary anymore. Next to this, another possible minor burden is 1 extra visit in addition to standard care.

ELIGIBILITY:
Inclusion criteria:

* Confirmed asthma diagnoses (≥12% and >200 ml reversibility in FEV1 or positive histamine/methacholine provocation test or FeNO ≥50) according to the asthma guidelines
* Diagnosed with severe, refractory asthma with eligibility for treatment with specific asthma biologics (omalizumab, mepolizumab, benralizumab, reslizumab, dupilumab) as determined at the regional asthma MDTM according to the asthma guidelines
* Age ≥ 18 years.
* Previous prescribed asthma biologics have to be ceased ≥ 4 times the half-life of that specific biologic.
* The patient has be relatively stable. The onset of an asthma exacerbation and/or a respiratory infection has to be ≥ 4 weeks ago.

Exclusion criteria:

* Primary COPD diagnosis.
* History of cancer:

  * Current basal cell carcinoma, localized squamous cell carcinoma of the skin or in situ carcinoma of the cervix. Patients are eligible to participate in the study provided that curative therapy was completed at least 12 months prior to the start of the study.
  * Current other malignancies. Patients are eligible to participate in the study provided that curative therapy was completed at least 5 years prior to the start of the study.
* Inability to sufficiently understand and read the Dutch language.
* Being unable to engage in a remote monitoring and coaching program through the use of a smartphone.
* Being unable to engage in physical activity (e.g. physical disability).
* Current pregnancy.
* Current breastfeeding.
* A liaison with the coordinating or (principal) investigator, which could likely influence the decision to participate in this study voluntarily (in concordance with the WMO - article 5).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Difference in percentage of patients treated with biologicals after 6 months of follow up | 6 months
  Difference in number of patients who receive treatment with biologics in the intervention arm compared with the control arm

SECONDARY OUTCOMES:
Difference in percentage of patients treated with biologicals after 12 months of follow up | 12 months
  Difference in number of patients who receive treatment with biologics in the intervention arm compared with the control arm
Difference in change in asthma control over time between the intervention- and control group | 6-12 months
  Asthma Controle assessed with the Asthma Control Questionnaire (ACQ-5). This questionnaire consists of five questions about the severity of symptoms which a patient experieces. The score range per question is 0-7 (0 = never and 7 = always). The total score will be calculated by dividing the sum of all scores by the amount of questions. A higher score is associated with worse asthma control.
Difference in change in quality of life over time between the intervention- and control group | 6-12 months
  Disease specific quality of life is measured with the Asthma Quality of Life Questionnaire (mini AQLQ). The mini AQLQ consists of 15 questions, which are subdivided into 4 domains (symptoms, activity limitation, emotional function and environmental stimuli). Each question has a 7-point scale (7 = not impaired at all - 1 = severely impaired). The overall score is the mean of all 15 responses. A lower score corresponds to a better quality of life.
Difference in asthma exacerbation frequency | 6-12 months
  Asthma exacerbation frequency

OTHER OUTCOMES:
Difference in change in spirometry and FeNO over time between the intervention - and control group. | 6-12 months
  Spirometry (e.g. FEV1, FVC) and FeNO measurements
Difference in direct healthcare consumption between the intervention- and control group | 6-12 months
  A Health Care Resource Utilization analysis will be performed by measuring the number of hospitalizations, the duration of hospitalization, the number of unscheduled visits to a health care provider (such as visits to the emergency department, general practitioner and outpatient clinic) all related to asthma and asthma exacerbations for which prednisolone with or without antibiotics was needed. This together with the cost of asthma biologics and equipment, staff and logistics for implementation and evaluation of EXACT@home.
Difference in prednisolone courses between the intervention- and control group. | 6-12 months
  Number of prednisolon courses
Difference in reduction in prednisolone maintenance therapy (if applicable) between the intervention and control group | 6-12 months
  Reduction in prednisolon maintenace therapy between the intervention- and control group. Reduction is defined as a decrease in prednisolon maintance therapy of ≥ 5 mg.
Difference in cumulative prednisolon dosage between the intervention- and control group. | 6-12 months
  Cumulative prednisolon dosage. The cumulative prednisolon dosage is the total amount of prednisolon a patient recieved during the year the patient participated in the study. The is calculated with prednisolone maintance therapy and prednisolone courses.
Difference in self-management between the intervention- and control group. | 6-12 months
  Knowledge, skills and confidence in being able to manage one's own health or illness: Patient Activation Measure (PAM). PAM is a questionnaire that measures knowledge, skills and trust in the ability to manage health or disease. The aim of PAM is to gain insight in the ability of the patient to improve their health status. It contains 13 questions that are rated on a 5-point scale. Based on the total score patients are scored along 4 levels: from very passive, not able to take control of their disease (PAM 1) towards active patients that feel completely in control of their disease (PAM 4).
Difference in dyspnea perception between the intervention- and control group. | 6-12 months
  Dyspnea perception is measured with the modified Medical Research Council (mMRC) dyspnea questionnaire. The MCR is a dyspnea scale, as a measure of disability in patients with respiratory disabilities. It consists of one question about shortness of breath and six possible answers. The score range 0 to 4 (0 = no shortness of breath at all and 4 = too breathless to leave the house or breathless with dressing/undressing). A higher score is therefore associated with a high burden of disease.
Difference in wellbeing between the intervention- and control group | 6-12 months
  Wellbeing is measured with the Wellbeing Of Older People (WOOP) questionnaire. The WOOP is a questionnaire which captures aspects relevant to the well-being of people. It consists of 9 questions. The scoring range for each question is from 1 to 5 (1 = no problems - 5 = very serious problems). The item scores will be summed to calculated the total score, which can range from 9 to 45, with higher scores indicating higher well-being.
Difference in patient satisfaction between the intervention- and control group | 6-12 months
  Patient satisfaction is measured with the Patients Assessment Chronic Illness Care (PACIC) questionnaire. The PACIC questionnaire measures specific actions or qualities of care, that patients report they have experienced in the delivery system. The survey includes 20 items, each with a score from 1 to 5 (1 = none of the time - 5 = always). The overall score is the mean of all 20 scores. The 20 items can also be divided into 5 subscales of which the mean can be calculated per subscale.
Measuring the change over time in physical activity in the intervention group | 6-12 months
  Physical activity (e.g. steps, percentage activity type) is measured with two activity trackers: the DynaPort Movemonitor from McRoberts and the Cardiowatch from Corsano.
Measuring the change over time in adherence and inhaler technique in the intervention group and the control group seperately | 6-12 months
  Adherence and inhaler technique are measured with the BF-Digihaler-DS, a digital inhaler which measures the moment of inhalation and inspiratory flow. Adherence is also measured with the Test of Adherence to Inhalers (TAI) questionnaire. TAI is a questionnaire which identifies patients with low adherence, determines the degree of adherence and gives an idea of the type or pattern of non-compliance. The TAI-10 consists of 10 questions and identifies patients with poor adherence and their degree of adherence. The scoring for each question ranges from 1 to 5 (1 = worst compliance - 5 = best compliance). All items provide a total score of between 10 (minimum) and 50 (maximum). A higher score is related to better adherence.
Observing sleeping patterns in the intervention group | 6-12 months
  Sleep is measured with the Cardiowatch from Corsano.
Observing vital parameters in the intervention group. | 6-12 months
  Vital parameters consists of the heart rate, respiratory rate, temperature. These are measured with the Cardiowatch from Corsano.
Measuring the differences in VOCs in exhaled breath measured with the eNose between baseline and follow-up in the intervention and in the control group separately. | 6-12 months
  VOCs in exhaled breath are measured with the Electronic Nose (eNose) from Breathomics
Monitoring of safety of the Digital inhaler (BF-Digihaler-DS from Teva) and eNose (Spironose from Breathomix). | 6-12 months
  Safety is measured by reporting adverse (device) events.
Monitoring and recording the course of treatment of each patient including the explanation behind changes in treatment (e.g. stopping treatment with biologicals). | 6-12 months
  The course of the treatment is documented for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: J.C.C.M. In 't Veen, dr., Principal Investigator — Franciscus Gasthuis & Vlietland
Locations (1):
- Franciscus Gasthuis & Vlietland, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bult L, Braunstahl GJ, Aerts JGJV, Banffer D, van Campen JSJA, van Daalen MS, van Dooren Y, Flanders U, Geurts ES, Hekking PP, Heller-Baan R, Jans MJA, Kappen JH, Mies RCA, Oppedijk B, de la Roij-Hartmans M, Van der Sar-Van der Brugge S, Turk Y, Vis E, Wolters R, Vasbinder EC, Veen JCCMI'. The effect of a systematic multi-dimensional assessment in severe uncontrolled asthma: a literature review and protocol for an investigator-initiated, open-label, randomized-controlled trial (EXACT@home study). BMC Pulm Med. 2025 May 17;25(1):240. doi: 10.1186/s12890-025-03646-5. PMID 40382637